CLINICAL TRIAL: NCT01489839
Title: Biomarkers of Periodontal Disease Progression
Status: Completed | Type: Observational
Sponsor: The Forsyth Institute (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); NYU Langone Health (Other); State University of New York at Buffalo (Other); University of Michigan (Other); Southern Illinois University (Other)
Responsible Party: Sponsor
Other Study IDs: 10-174-E; 5U01DE021127-02 (NIH)
Record Dates: First submitted 2011-12-06; First posted 2011-12-12 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2016-06

CONDITIONS: Periodontal Disease
Keywords: periodontal disease; biomarkers; periodontal treatment; clinical attachment level
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biological samples listed below will be obtained at baseline, each 2-month assessment visit for 12 months, and the 6-month post-therapy visit.
  Blood. Ten mL of blood will be obtained by venipuncture from the antecubital fossa. Subjects consenting to have a blood sample drawn for future DNA analysis will have an additional 7 mL of blood drawn at the baseline visit.
  Saliva. Each subject will provide a timed sample of whole saliva by expectorating into a sterile graduated cylinder.
  Gingival crevicular fluid. A GCF sample will be collected from the mesial and distal aspect of each posterior tooth (excluding third molars) using filter strips (Periopaper®) gently inserted 1 to 2 mm subgingivally. A total of up to 32 samples will be obtained.
  Subgingival plaque samples. Two plaque samples will be taken from the mesial and distal aspects of each posterior tooth (excluding third molars) for up to 64 samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Periodontal diseased: Subjects with periodontal disease will be enrolled. Subjects with mild disease will have at least 4 teeth with at least 1 site with pocketing of 5 mm or more and concomitant attachment greater than or equal to 2 mm, and radiographic evidence of mesial or distal alveolar bone loss around at least 2 of the affected teeth. Subjects with severe disease will have at least 8 teeth with a site having >5mm pocketing and loss of 3 mm attachment with evidence of alveolar bone loss in 2 teeth.
  Interventions: Other: Periodontal therapy
- Periodontally healthy: Periodontally healthy subjects have no teeth with pocketing of 4 mm or greater and attachment loss, with the exception of the distal of the second molars where a pocket of 4 mm and concomitant attachment of up to 2 mm will be acceptable. Healthy subjects can have up to 3 sites with gingival recession and no radiographic evidence of alveolar bone loss.
  Interventions: Other: Periodontal therapy

INTERVENTIONS:
Other: Periodontal therapy — All subjects will have professional dental prophylaxis and periodontal therapy withheld for 12 months during the disease progression and monitoring phase. After 12 months, subjects with periodontal disease will receive periodontal therapy to consist of scaling and root planing, and periodontally healthy subjects will receive professional dental prophylaxis. Subjects with periodontal disease will also receive Supportive Periodontal Therapy at the 3- and 6-month post-therapy visits. Subjects showing periodontal disease progression greater than a predetermined threshold during the monitoring or maintenance phases of the study will be given rescue therapy consisting of placement of a local antibiotic at the site of disease progression.

SUMMARY:
The primary purpose of the study will be to look for biological biomarkers to determine which people with gum disease will have a worsening of the disease. A second objective of this study will be to look at the effects of periodontal treatment on the levels of the biomarkers that are identified.

DETAILED DESCRIPTION:
This multicenter clinical study will investigate biomarkers of periodontal disease progression. The study will enroll 375 subjects with periodontal disease and 125 periodontally healthy subjects. All subjects will be monitored clinically and have samples taken every 2 months for 12 months for analysis of inflammatory and immunological biomarkers and microbial species. Subjects displaying periodontal disease progression greater than an established threshold will receive periodontal rescue therapy at progressing periodontal sites and continue with monitoring. Periodontally healthy subjects and non-progressing sites in subjects with periodontal disease will serve as controls. After 12 months, subjects with periodontal disease will receive periodontal therapy consisting of 4 quadrants of scaling and root planing. Periodontally healthy subjects will receive prophylaxis and scaling and exit the study. Following periodontal therapy, subjects with periodontal disease will be followed for a maintenance period of 6 months for clinical and biological monitoring. Statistical analyses will compare biomarkers and microbial species between periodontally healthy subjects and subjects with periodontal disease, between progressing and non-progressing periodontally diseased sites, and between periodontally diseased sites before and after periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

To be eligible to participate in this study, a subject must meet all of the following criteria:

1. Ability to understand, and willingness and ability to read and sign, the informed consent form.
2. Age of at least 25 years.
3. Ability to understand and follow directions for study procedures.
4. Minimum of 20 natural teeth, excluding third molar teeth; at least 12 of these teeth must be pre-molars, first molars, or second molars.
5. Willingness not to have professional dental prophylaxis or scaling for the duration of the disease progression and monitoring phase (12 months).
6. Willingness to comply with all study procedures and be available for the duration of the study.
7. For women with reproductive potential, willingness to use highly effective contraception (e.g., licensed hormonal contraception, intrauterine device, abstinence, or vasectomy in partner).

Specific inclusion criteria:

Healthy periodontal subjects must have:

1. Any tooth with 3 mm or less PD, irrespective of the attachment level, will be acceptable
2. No teeth with PD of 4 mm or more and concomitant attachment loss, with the exception of the distal of the second molars where a PD of 4 mm and concomitant CAL of up to 2 mm will be acceptable.
3. No radiographic evidence of alveolar bone loss (defined as a distance of greater than 2.0 mm measured radiographically from the CEJ to the crest of the alveolar bone); with the exception of the mandibular incisors where up to 3.0 mm of alveolar bone loss measured radiographically from the CEJ to the crest of the alveolar bone will be accepted.

Mild periodontal disease subject: periodontal loss must meet the following criteria and must not meet the minimum criteria for severe periodontal loss:

1. At least 4 teeth with at least 1 site of PD of 5 mm or more and concomitant CAL greater than or equal to 2 mm, and radiographic evidence of mesial or distal alveolar bone loss around at least 2 of the affected teeth. Alveolar bone loss is defined as a distance of > 2.0 mm measured radiographically from the CEJ to the crest of the alveolar bone.

Subjects with severe periodontal loss must meet all of the following criteria:

1. At least 8 separate teeth with at least 1 site of PD of 5 mm or more and concomitant CAL greater than or equal to 3 mm, and radiographic evidence of mesial or distal alveolar bone loss around at least 2 of the affected teeth. Alveolar bone loss is defined as a distance of > 2.0 mm measured radiographically from the CEJ to the crest of the alveolar bone.

Exclusion Criteria:

1. Presence of orthodontic appliances.
2. The following conditions noted on oral examination:

   * Oral lichen planus
   * Candidiasis
   * Clinical leukoplakia
   * Clinical erythroplakia
   * Pemphigus
   * Pemphigoid
   * Other recurrent intraoral or perioral vesiculobullous diseases
   * Aphthous ulcerations (major or minor). Subjects presenting with aphthous ulcers should be rescreened after 2 weeks. They will be eligible if the ulcers have healed and the subject does not have a history of frequent recurrences.
   * Herpetic lesions. Subjects presenting with herpes labialis or intraoral herpes should be rescreened after 2 weeks. They will be eligible if the lesions have healed and the subject does not have a history of frequent recurrences.

     j. Traumatic ulcers. If a subject presents with a traumatic ulcer, he/she can be rescreened in 2-3 weeks. The subject will be eligible if the ulcers have healed.
3. Acute necrotizing ulcerative gingivitis or gross tooth decay, as determined by the investigator.
4. Root fragments, pericoronitis, endo-perio lesions, or other dental abscesses. Subjects may be rescreened after resolution of these dental conditions.
5. Pregnancy or lactation.
6. Requirement for prophylactic antibiotics for dental procedures (e.g., for certain heart and orthopaedic conditions*).
7. Periodontal or systemic antibiotic therapy in the previous 6 months. Routine dental prophylaxis will be allowed.
8. Use of cigarettes or other tobacco products within 1 year before the screening visit.
9. Any medical condition that might influence the course of periodontal disease or treatment (e.g., diabetes [irrespective of level of control], human immunodeficiency virus infection or acquired immunodeficiency syndrome, use of medications associated with gingival hyperplasia).
10. Chronic use of nonsteroidal anti-inflammatory drugs (e.g., for arthritis), defined as the need, or anticipated need, for over 3 weeks of continuous use at the time of enrollment or during the course of the study. The use of low-dose aspirin (81 mg/day) for prophylaxis will be allowed.
11. Current or anticipated use of chronic systemic corticosteroids, cyclosporine, or other systemic immunosuppressive agent. The use of inhaled corticosteroids will be allowed.
12. Hypersensitivity to tetracyclines (e.g., tetracycline, doxycycline, minocycline).
13. Participation in a clinical study testing a drug, biologic, device, or other intervention within the last 30 days.
14. Any condition or circumstance that, in the opinion of the investigator, would place the subject at increased risk or preclude his/her full compliance with or completion of the study.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 500 subjects (375 subjects with periodontal disease and 125 periodontally healthy subjects) will be enrolled at 4 centers in the US.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2012-01; Primary Completion 2016-06 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Attachment Level (CAL) | After the baseline visit, subjects will return to the clinic every 2 months (± 7 days relative to baseline) for 12 months.
  The primary study outcome will be progression of periodontal disease as determined by CAL. Initial disease progression at a site will be defined as loss of ≥2 mm in CAL at any assessment or follow-up visit compared with baseline. Subsequent disease progression will be similarly defined except that the loss in CAL will be compared with the last visit at which disease progression was detected.

SECONDARY OUTCOMES:
Biomarker Levels compared between progressing and non-progressing sites as determined by CAL changes | Levels measured every 2 months for 12 months
  Biomarker levels will be compared between progressing and non-progressing periodontally diseased sites. The biomarkers include microbial species in saliva, GCF, and plaque and inflammatory and immunological markers in serum, saliva, and GCF. In addition, differences will be compared between diseased subjects before and after periodontal therapy and between periodontally diseased and healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo P Teles, DDS, DMSc, Principal Investigator — The Forsyth Institute
Locations (5):
- United States (5):
  - Southern Illinois University, Edwardsville, Illinois
  - The Forsyth Institute, Cambridge, Massachusetts
  - University of Michigan School of Dentistry, Ann Arbor, Michigan
  - State University of New York at Buffalo, Buffalo, New York
  - NYU College of Dentistry, New York, New York

REFERENCES:
- [Derived] Yost S, Duran-Pinedo AE, Teles R, Krishnan K, Frias-Lopez J. Functional signatures of oral dysbiosis during periodontitis progression revealed by microbial metatranscriptome analysis. Genome Med. 2015 Apr 27;7(1):27. doi: 10.1186/s13073-015-0153-3. eCollection 2015. PMID 25918553